CLINICAL TRIAL: NCT03070028
Title: Randomized Prospective Comparison of Crystallized Phenol and Platelet Rich Plasma Applications in Treatment of Pilonidal Sinus Disease
Brief Title: Minimally Invasive Treatment Methods for Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Barış Sevinç, assistant proffessor, Uşak University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PS001
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenol (Experimental): crystallised phenol application
  Interventions: Procedure: crystallised phenol
- platelet rich plasma (Experimental): PRP application
  Interventions: Procedure: Platelet rich plasma

INTERVENTIONS:
Procedure: crystallised phenol — crystallised phenol will be applied to sinus cavity
  Arms: Phenol
Procedure: Platelet rich plasma — platelet rich plasma will be applied to sinus cavity
  Arms: platelet rich plasma

SUMMARY:
Patients with pilonidal sinus disease will be randomised to two groups (crystallised phenol and platelet rich plasma). Sinus healing time, patient satisfaction, complications and recurrence rates will be compared.

DETAILED DESCRIPTION:
Patients with pilonidal sinus disease will be treated by either crystallised phenol or platelet rich plasma application. Treatment results, healing time, postprocedural complications, patient satisfaction and recurrences will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Having pilonidal sinus disease
* accepting to be involved in the study

Exclusion Criteria:

* below the age of 18
* having connective tissue disorders
* diabetes mellitus
* severe anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
healing time | first 1 year of the study
  Time to complete closure of the sinus cavity.

CONTACTS AND LOCATIONS:
Overall Officials: Barış Sevinç, M.D., Principal Investigator — Uşak University Medical School
Locations (1):
- Uşak University, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sevinc B, Damburaci N, Karahan O. Comparison of Curettage Plus Platelet-Rich Plasma Gel and Curettage Plus Phenol Application in Treatment of Pilonidal Sinus Disease: A Randomized Trial. Dis Colon Rectum. 2022 May 1;65(5):735-741. doi: 10.1097/DCR.0000000000002082. PMID 34629430